CLINICAL TRIAL: NCT06793176
Title: Diagnostic Accuracy of Vibraimage Technology for Detecting Depression in a Psychiatric Outpatient Setting
Brief Title: Vibraimage Technology for Detecting Depression in Psychiatric Outpatients
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing HuiLongGuan Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Professor, Peking University People's Hospital
Other Study IDs: Vibraimage_Psychiatric
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Depressed Group: This group consists of individuals who were ultimately diagnosed with depression by a specialist physician.
  Interventions: Diagnostic Test: Video capture
- Non-Depressed Group: This group consists of individuals who were ultimately diagnosed as not having depression by a specialist physician.
  Interventions: Diagnostic Test: Video capture

INTERVENTIONS:
Diagnostic Test: Video capture — A 20-second video capture of head-neck movements at high frame rates is conducted for all participants to obtain high-resolution images. The captured videos are analyzed using an algorithm based on Vibraimage technology to infer whether the participants have depression.

SUMMARY:
Vibraimage technology captures high-frame-rate images of head-neck movements, converting them into vibraimages that display muscle vibration amplitude and frequency. Using algorithms and calculations, it derives an emotional index from these images. This non-contact, objective method analyzes psychological indicators through micro-movement detection. An algorithm has been developed to detect depression by calculating 12 emotional and 2 psychophysiological parameters. This diagnostic accuracy study aims to validate the technology's ability to diagnose depression in psychiatric outpatients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 70 years.
* No difficulties in reading or writing Chinese; fluent in Mandarin.
* Currently not taking psychotropic medications or on a stable dose for at least 6 weeks.
* Provided informed consent to participate in the study.

Exclusion Criteria:

* Schizophrenia.
* Bipolar disorder.
* History of organic brain disease or significant head trauma.
* Presence of severe systemic medical conditions.
* Suicidal ideation or a score ≥3 on Item 3 ("Suicide") of the 17-item Hamilton Depression Rating Scale (HAMD-17).
* Substance dependence or abuse.
* Intellectual disability or dementia.
* Inability to complete video capture or cooperate due to uncontrollable factors (e.g., hyperactivity, Parkinson's disease, or other conditions that prevent remaining still)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Psychiatric outpatients attending the Beijing Huilongguan Hospital during the study period.
Sampling Method: Probability Sample
Enrollment: 601 (Actual)
Dates: Start 2025-01-26 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
discrimination | Participants undergo video capture and same-day clinical diagnosis by a physician. Video analysis and suggestive diagnosis are completed on the following day.
  The primary outcome measure is the diagnostic discrimination of Vibraimage technology for depression, assessed by calculating the area under the receiver operating characteristic (ROC) curve. Participants first undergo video capture, followed by a clinical diagnosis of depression by a physician. Both the physician and participants are blinded to the results of the video analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing HuiLongGuan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available to qualified researchers upon reasonable request. Data sharing will be subject to approval by the principal investigator (PI) and the study sponsor.

REFERENCES:
- [Derived] Jiang B, Zhang Y, Xie Z, Wu Z, Ma Y, Zhang X, Feng Y. A novel non-contact screening tool based on Vibraimage technology for detecting depressive disorder in psychiatric outpatients: A diagnostic accuracy study. J Affect Disord. 2026 Jan 1;392:120232. doi: 10.1016/j.jad.2025.120232. Epub 2025 Sep 2. PMID 40907713